CLINICAL TRIAL: NCT06946017
Title: Effect of a Fermented Whey and Fiber Supplement on Digestive Comfort of Recreational Athletes With and Without GI Complaints
Brief Title: Effect of a Fermented Dairy Protein With Prebiotic Fiber on GI Complaints
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Friesland Campina (Unknown)
Responsible Party: Principal Investigator, Floris Wardenaar, Assistant Professor in Nutrition, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: STUDY00020575
Record Dates: First submitted 2025-04-17; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Digestive Health; Quality of Life
Keywords: Participants; Healthy subjects; Athlete; Women; Men; Fermented Dairy; Prebiotics; Gut microbiota; Self-reported; GI-tract; Diet; Immune markers; Exercise
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Motor Activity

STUDY DESIGN:
Intervention Model Description: Part I is a crossover design. Part II is a parallel design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented dairy protein with prebiotic fiber (Experimental): During 3-week period participants consume a fermented dairy protein with prebiotic fiber.
  During Part I participants are randomly assigned to start with the experimental arm or the control arm, after a 3-week washout period, they will supplement again for 3 weeks with the opposite supplement (double blind, randomized cross-over trial).
  During Part II participants are randomly assigned to the experimental arm only (double blind, randomized parallel trial).
  Interventions: Dietary Supplement: Fermented dairy protein with prebiotic fiber supplement
- Control protein supplement (Placebo Comparator): During 3-week period participants consume a control supplement.
  During Part I participants are randomly assigned to start with the control arm or the experimental arm, after a 3-week washout period, they will supplement again for 3 weeks with the opposite supplement (double blind, randomized cross-over trial).
  During Part II participants are randomly assigned to the control arm only (double blind, randomized parallel trial).
  Interventions: Dietary Supplement: Control placebo

INTERVENTIONS:
Dietary Supplement: Fermented dairy protein with prebiotic fiber supplement — Both the intervention and placebo products contain a serving of 15g with ~53Kcal, 0.5g Fats, 5g Carbohydrate, 7.5g Protein that need to be dissolved as powder in water in a protein shaker that will be provided. The intervention product contains whey protein concentrate and a prebiotic fiber. All ingredients that are designated by the FDA as Generally Recognized as Safe (GRAS). Participants will be asked to take the supplement daily before breakfast.
  Arms: Fermented dairy protein with prebiotic fiber
Dietary Supplement: Control placebo — Both the intervention and placebo products contain a serving of 15g with ~53Kcal, 0.5g Fats, 5g Carbohydrate, 7.5g Protein that need to be dissolved as powder in water in a protein shaker that will be provided. The placebo product is calorically matched to the intervention product and the main ingredients are protein and carbohydrate. All ingredients that are designated by the FDA as Generally Recognized as Safe (GRAS). Participants will be asked to take the supplement daily before breakfast.
  Arms: Control protein supplement

SUMMARY:
A positive impact of a fermented dairy protein with prebiotic fiber supplement on self-reported GI complaints and wellbeing has been suggested (Wardenaar et al. 2024). The following project aims to further investigate the impact of this supplements in athletes with and without GI complaints in two separate data collections.

Part I of the data collection aims to investigate the impact of this supplement vs. a placebo on carbohydrate malabsorption (as a potential cause for GI distress) in athletes that normally don't identify as having GI complaints (randomized double-blind cross over study design covering a total of 9 weeks, including a 3-week washout period).

Part II of the data collection aims to confirm the earlier found results in the previous study (Wardenaar et al. 2024) in a group athletes self-reporting GI complaints that will be randomized into an intervention group or a placebo group (randomized double-blind parallel study design covering a total of 3 weeks).

DETAILED DESCRIPTION:
A substantial number of athletes suffer from gastro-intestinal (GI) problems, which may impair performance and/or subsequent recovery. Regardless of the prevalence of GI complaints, gut barrier integrity is impaired with high-intensity training. Emerging studies show a positive correlation between the gut microbiome and GI problems and general health and wellbeing.

This project will perform two well-controlled studies:

Part I will be looking into the impact of a 3-week supplementation of fermented dairy protein with prebiotic fiber supplement vs. 3-week supplementation of a control supplement on carbohydrate malabsorption (by means of a lactose tolerance test), Bifidobacterium, GI complaints, general well-being and overall gut microbiota in people screened for not reporting substantial GI complaints while being lactose non-persistent (LNP) and/or being responsive to a lactose tolerance test.

Part II investigates the impact of a 3-week supplementation of a fermented dairy protein with prebiotic fiber supplement vs. a control supplement on GI complaints, Bifidobacterium, general well-being, overall gut microbiota, immune markers, gut redox status, and short chain fatty acids in feces in people screened for reporting substantial GI complaints.

Both study parts include multiple standardized exercise tests before and after each supplementation period (Part I: 4 exercise testing days, Part II: 2 exercise testing days). The participants will come in fasted (after not eating starting 10 pm the night before) and they will perform a 60-minute hiking protocol in a warm environment. After the first-time participants will copy their personal exercise protocol during the following session(s). The exercise exists of hiking on a treadmill in a warm environment (30-35°C), while reaching an exercise intensity of 70% of the subject's VO2 max. Which is an intensity in which the subject has an elevated breathing frequency but is still able to talk.

SCREENING After being eligible on paper (based on the results of an online screening questionnaire) people are invited to sign informed consent via REDCap, a secure, web-based application designed for building and managing online surveys and databases for research studies.

For Part I an addition screening step is included to determine eligibility, including a buccal swab to determine lactose non-persistence (to identify the CC gene), as well as a lactose tolerance test (administration of a dose of 25g of lactose mixed into 250mL, with hydrogen breath measurements at 30-, 60- and 90-minutes after lactose consumption). For Part II no additional screening will be performed.

FAMILIARIZATION VISIT Before performing any exercise, body height and weight, as well as waist and hip circumference will be taken by a research team member, and some additional questions will be asked about exercise and diet habits. After this the participant will perform a maximal exercise test, that will be used to determine the exercise intensity during the following exercise sessions. For this purpose, the Balke protocol will be used and VO2 max will be measured. This test includes a treadmill walking/hiking test including progressive stages where the incline increases each minute (by 1%), but the speed remains 3.3mph.

EXERCISE TEST (PART I and PART II) The treadmill will start at 70% of the final incline determined by the max test and participants will start the speed determined by the familiarization test and will be increased as necessary to achieve a heart rate associated with 70% of the VO2max measured during the familiarization visit using a Balke test. Heart rate and speed will be continuously monitored, when speed needs to be adjusted at a later phase during the protocol (because heart rate is not within the targeted HR-range), this will be registered to allow for exact copying the protocol during the next exercise sessions. The exercise will consist of 60 minutes of steady-state exercise. A rating of perceived exertion (RPE) measure via a BORG visual analog scale will be taken every 10-minutes to ensure participants are maintaining a moderate level activity. Only during Part I participants will receive a feeding after the exercise test. Participants will receive at the end of the exercise test 25g lactose mixed into 250mL water, no food will be provided after the heat stress test, but water can be consumed ad libitum.

PART I This part has a randomized controlled cross-over design: Some of the data collection will take place at home (e.g the collection of stool samples, 1-3 minutes per sample, 4-12 minutes total, and filling out a GSRS questionnaire the day after each exercise test for 1-3 minutes per questionnaire, 4-12 minutes total), as well as the consumption of the intervention product or placebo (1-2 minutes per day, 21-42 minutes total), but the majority of the measurements will be collected at our research facility.

Measurements for different testing days for Part I:

Day ≤0: Screening questionnaire (allowing to select eligible athletes based on the criteria listed in inclusion and exclusion criteria). Sign informed consent, perform exercise test to determine heart rate submax including measuring body composition. Provide instructions and provide stool sample collection materials.

Test Day 0, 21, 42, 63: Fecal swab (for microbiota-redox activity) before arrival; Self-reported digestive comfort, general wellbeing (PHQ. K6, SVS), and dietary questionnaires at arrival. Blood sample is taken based on a finger prick using a lancet method (for SCFA/LBP) before the exercise test followed by the exercise test, and another finger prick (~150 uL blood for LBP). After the lactose dose is consumed post-exercise, multiple hydrogen breath samples are collected (malabsorption). Hydrogen measurements will be issued at baseline (-60 min), post-exercise (0 min), 30-minutes post-exercise (30 min), 60-minutes post-exercise (60 min), 90-minutes post-exercise (90min), 120-minutes post-exercise (120min) 150-minutes post-exercise (150min), 180-minutes post-exercise (180min), 210-minutes post exercise and 240-minutes post exercise (240min). Hydrogen breath analysis is a minimally invasive procedure which requires the participant to breath normally but exhale into a gas sample bag until the 250mL bag is filled. Prior to taking a hydrogen breath sample, a 10mL mouthwash rinse followed by a rinse with water to prevent bacterial flora from affecting the hydrogen breath measures will be completed before each measure of hydrogen.

Accompanying the hydrogen breath test at 0 min, 60 min, 120 min, 180 min and 240 min, an adjusted GSRS questionnaire will also be given for self-reported digestive comfort during the last 60 minutes.

Test Day 0+1; Day 21+1, Day 42+1, Day 63+1: Before the exercise stress test the regular GSRS will be provided to reflect self-reported digestive comfort during the last week, and a 24-hour after exercise an adjusted GSRS questionnaire will be provided to assess the last 24-h for self-reported digestive comfort.

Research questions for Part I:

Question 1: For Part I: Does 3-week supplementation of a fermented dairy protein with prebiotic fiber supplement lowers lactose malabsorption reflected by consecutive hydrogen breath measurements compared to a control after 60-minute hiking exercise in the heat.

Question 2: For Part I: Does 3-week supplementation of a fermented dairy protein with prebiotic fiber supplement increase fecal Bifidobacterium compared to a control.

Question 3: For Part I: Does 3-week supplementation of a fermented dairy protein with prebiotic fiber supplement result in positive changes in GI complaints based on a modified gastro-intestinal symptom rating scale (GSRS) during the lactose tolerance test after 60-minute hiking exercise in the heat.

Question 4: For Part I: Does 3-week supplementation of a fermented dairy protein with prebiotic fiber supplement result in positive changes in general wellbeing (measured via multiple questionnaires) and general gut microbiota.

PART II This part has a randomized controlled parallel design: Some of the data collection will take place at home (e.g the collection of stool samples, 3-6 minutes for two samples a time, 6-12 minutes total, and filling out a GSRS questionnaire the day after each exercise test for 1-3 minutes per questionnaire, 2-6 minutes total), as well as the consumption of the intervention product or placebo (1-2 minutes per day, 21-42 minutes total), but the majority of the measurements will be collected at our research facility.

Measurements for different testing days for Part II:

Screening (Day ≤0): Screening questionnaire (select eligible athletes based on inclusion and exclusion criteria); Sign informed consent, perform exercise test to determine heart rate submax, including measuring body composition. Provide instructions and provide stool sample collection materials.

Baseline (Day 0) and Endpoint (Day 21): Fecal swab (for microbiota-redox activity, SFCA composition) before arrival; Venous blood sample (5 mL to measure TNF-a, CRP, IL-4, IL-6, IL-8, IL-10, MCP-1) and saliva (check swab to measure sIgA, and assessment of flow rate) collection for immune markers; Self-reported digestive comfort, general wellbeing (PHQ. K6, SVS), and dietary questionnaires filled out online. An additional blood sample is taken based on a finger prick using a lancet method (~250 uL blood to measure SCFA and LBP) before the exercise test followed by the exercise test, and another finger prick (to measure LBP again).

Day 0+1 and Day 21+1: day after exercise stress test: A 24-hour after exercise adjusted GSRS questionnaire will be provided to assess the last 24-h for self-reported digestive comfort.

Research questions for Part II:

Question 5: For Part II: Does 3-week supplementation of a fermented dairy protein with prebiotic fiber supplement lowers GI complaints based on a modified gastro-intestinal symptom rating scale (GSRS) before, directly after, and 24-hours after 60-minute hiking exercise in the heat compared to a control.

Question 6: For Part II: Does 3-week supplementation of a fermented dairy protein with prebiotic fiber supplement increase fecal Bifidobacterium compared to a control.

Question 7: For Part II: Does 3-week supplementation of a fermented dairy protein with prebiotic fiber supplement result in positive changes in general wellbeing (measured via multiple questionnaires) and general gut microbiota compared to a control.

Question 8: For Part II: Does 3-week supplementation of a fermented dairy protein with prebiotic fiber supplement result in positive changes in immune markers, gut redox status and fecal short chain fatty acids compared to a control.

ELIGIBILITY:
Aside from having participants fitting the inclusion and exclusion criteria below, potential participants will be screened using the gastrointestinal symptom rating scale (GSRS). Based on the outcome they will be assigned to the Part I (i.e. no self-reported GI tract issues (GSRS questionnaire score GI complaints, based on GSRS screening with all items scored <4 (severe) and a total GSRS score ≤25), or Part II (i.e. Severe self-reported GI tract issues (GSRS questionnaire score GI complaints, based on GSRS screening with at least one item scored ≥4 (severe) and a total GSRS score ≥30). If they don't fit these criteria (i.e., having a GSRS score ranging from 26-29) they will be excluded from participation.

Inclusion Criteria:

* Healthy subjects living in the Phoenix area in AZ, USA during the study
* Women/Men aged between 18-50 years (50-50%)
* Recreational competitive and non-competitive athletes (exercise at least 2x per week with a minimal total duration of 2 hours/week)
* BMI value between ≥18.5 and ≤ 30 kg/m2
* No physical limitations due to an injury (i.e., able to perform all activities associated with daily living and exercise in an independent manner).
* Willing to slightly increase their energy intake via a supplement during the study period on daily basis in the morning before breakfast.
* Willing and comfortable to perform multiple physical (stress) tests on a treadmill during the study.
* Participants without any contraindications when scoring the Physical Activity Readiness Questionnaire (PAR-Q+).
* Written informed consent
* For part I: Self-perceived lactose intolerance, and/or omission of dairy products, and/or identifying as Hispanic/Latino or Asian
* For part I: Determined to be lactase non-persistent (LNP) CC genotype by qPCR, and/or positive lactose intolerance test (>20ppm increase from baseline when 25g of lactose administered)

Exclusion Criteria:

* Users of (sport) supplements containing probiotics and/or prebiotics and those unwilling to temporarily stop use of these supplements at least 3 weeks prior to start of the intervention
* Women who plan to start or stop the use of contraceptives before or during study period
* Women that have additional or worse GI symptoms during their period that can be classified as severe
* Smoking
* Clinical lactose intolerance
* Clinical or self-perceived milk protein allergy
* Diagnosed GI tract disorders or diseases
* Musculoskeletal disorders
* Diagnosed metabolic disorders (such as diabetes)
* Use of any medications known to affect protein metabolism (i.e., corticosteroids, non-steroidal anti-inflammatories, or prescribed acne medications).
* Chronic use of gastric acid suppressing medication or anti-coagulants
* Chronic use of anti-inflammatory medication
* Use of antibiotics the past 0-6 months
* Blood donation in the past 2 months
* (Intending to become) Pregnant/lactating women
* Significant changes in body weight during the past 4 weeks (i.e., due to reduction of body weight through limiting caloric intake, illness,)
* Athletes should not aim to lose bodyweight by reducing energy intake during the study
* For Part I: A hydrogen breath peak of less than 20 ppm over baseline during a lactose tolerance test

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Part I: Hydrogen in breath | For 240 minutes post exercise after consuming a bolus of lactose.
  Hydrogen in breath as indicator of lactose malabsorption.
Part II: Gastrointestinal Symptoms Rating Scores | For 240 minutes post exercise after consuming a bolus of lactose.
  Gastrointestinal Symptoms Rating Scores (GSRS) as indicator of self-reported digestive comfort. The GSRS is a 15-item self-administered questionnaire divided into five clusters of symptoms: reflux, abdominal pain, indigestion, diarrhea, and constipation. These symptoms are graded on a 7-point Likert scale, where 1 signifies no discomfort at all and 7 represents very severe discomfort. The total score will be calculated, as well as the percentage of subjects reporting symptoms (≥2), or moderate to severe symptoms (≥4). A minimal score of indicates no GI symptoms, whereas a score up to 105 suggests extreme GI symptoms.

SECONDARY OUTCOMES:
Part I and Part II: Fecal Bifidobacterium | Stool sample collected at least one day before the test day including the exercise test
  Fecal Bifidobacterium as a (partial) mechanistic explanation for a change in carbohydrate (lactose) absorption or self-reported digestive comfort.

OTHER OUTCOMES:
Part I: Gastrointestinal Symptoms Rating Scores | Covering the last 7 days before each testing day.
  Gastrointestinal Symptoms Rating Scores (GSRS) as indicator of self-reported digestive comfort. The GSRS is a 15-item self-administered questionnaire divided into five clusters of symptoms: reflux, abdominal pain, indigestion, diarrhea, and constipation. These symptoms are graded on a 7-point Likert scale, where 1 signifies no discomfort at all and 7 represents very severe discomfort. The total score will be calculated, as well as the percentage of subjects reporting symptoms (≥2), or moderate to severe symptoms (≥4). A minimal score of indicates no GI symptoms, whereas a score up to 105 suggests extreme GI symptoms.
Part I and Part II: Self-reported general wellbeing | At each testing day, before the exercise test.
  Self-reported general wellbeing using the Physical Health Questionnaire (PHQ). The PHQ covers sleep disturbance, headache, GI problems, and respiratory infections using 14 items with Likert scales scoring in the range of 1-7, from "not at all" to "all the time". The total score is in the range of 14-98, where a low score indicates better physical health.
Part I and Part II: Self-reported general wellbeing | At each testing day, before the exercise test.
  Self-reported general wellbeing using the psychological Distress Scale (K6). The K6 addresses depressed mood, motor agitation, fatigue, worthless guilt, and anxiety. The K6 uses a 0-3 Likert scale, ranging from "none of the time" to "all of the time". Total score is in the range of 0-18, where a low score indicates low mental distress, with ≥13 suggesting mental distress.
Part I and Part II: Self-reported general wellbeing | At each testing day, before the exercise test.
  Self-reported general wellbeing using the subjective vitality scale (SVS). The SVS holds 7 items covering feelings related to energy and feeling alive with Likert scales scoring in the range of 1-7, from "not at all true" to "very true". The total score is in the range of 7-49, where a low score indicates not being feeling vital and energized, whereas higher scores suggest the opposite.
Part I and Part II: Gut microbiota composition | Stool sample collected at least one day before the test day including the exercise test.
  Gut microbiota composition of fecal samples based on 16s microbial profiling.
Part I and Part II: Nutrient intake | At each testing day, within 240 minutes after the exercise test.
  Nutrient intake using ASA24 dietary recalls to report energy and macro- and micronutrient intake of the day before the exercise test.
Part I and Part II: Diet quality | At each testing day, after the exercise test
  Diet quality using REAP questionnaire covering food group consumption over the last 7 days before the exercise test
Part II: Immune markers | At each testing day, before the exercise test.
  Immune markers in blood (TNF-a, CRP, IL-4, IL-6, IL-8, IL-10, MCP-1) and saliva (IgA).
Part II: Short chain fatty acids | At each testing day, before the exercise test.
  Short chain fatty acids (SCFA) in fecal samples (absolute values for acetate, and relative abundance for the full SCFA panel).
Part II: Gut redox status | Stool sample collected at least one day before the test day including the exercise test.
  Gut redox status based on gut microbiota analysis
Part I and II: Gut integrity | Pre and post exercise on a testing day, within 5 minutes before and 5 minutes after the exercise test.
  Gut integrity based on LBP in blood.
Part I and II: Gastrointestinal Symptoms Rating Scores 24 after exercise | Covering the last 24 hours after the exercise test, the day after the exercise test.
  Gastrointestinal Symptoms Rating Scores (GSRS) as indicator of self-reported digestive comfort. The GSRS is a 15-item self-administered questionnaire divided into five clusters of symptoms: reflux, abdominal pain, indigestion, diarrhea, and constipation. These symptoms are graded on a 7-point Likert scale, where 1 signifies no discomfort at all and 7 represents very severe discomfort. The total score will be calculated, as well as the percentage of subjects reporting symptoms (≥2), or moderate to severe symptoms (≥4). A minimal score of indicates no GI symptoms, whereas a score up to 105 suggests extreme GI symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- ASU Health Futures Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
This is up to the industry funder to allow sharing.

REFERENCES:
- [Background] Wardenaar FC, Mohr AE, Ortega-Santos CP, Nyakayiru J, Kersch-Counet C, Chan Y, Clear AM, Kurka J, Schott KD, Seltzer RGN. Explorative Characterization of GI Complaints, General Physical and Mental Wellbeing, and Gut Microbiota in Trained Recreative and Competitive Athletes with or without Self-Reported Gastrointestinal Symptoms. Nutrients. 2024 May 30;16(11):1712. doi: 10.3390/nu16111712. PMID 38892645